CLINICAL TRIAL: NCT00419341
Title: A Phase III Open-Label, Prospective, Multicenter Study of the Efficacy, Tolerability, Safety, and Pharmacokinetics of Immune Globulin Subcutaneous (Human), IgPro20 in Subjects With Primary Immunodeficiency (PID)
Brief Title: Study of Subcutaneous Immunoglobulin in Patients With PID Requiring IgG Replacement Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB04_009CR; 1458 (Other: CSL Behring)
Record Dates: First submitted 2006-12-22; First posted 2007-01-08 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2012-12

CONDITIONS: Primary Immune Deficiency
Keywords: Immune globulin subcutaneous; SCIG; Primary immunodeficiency; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Hizentra

ARMS (1):
- IgPro20 (Experimental): Human Normal Immunoglobulin for Subcutaneous Administration (IgPro20) is a liquid formulation of normal human IgG at a concentration of 20% administered as a SC infusion at weekly intervals. The initial weekly dose was determined based on subjects' previous treatment. Dose adjustments could be performed during the wash-in/wash-out period at the discretion of the investigator.
  Interventions: Biological: Human Normal Immunoglobulin for Subcutaneous Administration

INTERVENTIONS:
Biological: Human Normal Immunoglobulin for Subcutaneous Administration
  Other Names: Hizentra

SUMMARY:
The objective of this study is to assess the efficacy, tolerability, safety and pharmacokinetics of IgPro20 in patients with primary humoral immunodeficiency (PID).

DETAILED DESCRIPTION:
The entire study consists of a 12-week wash-in/wash-out period followed by a 12-month treatment period. Pharmacokinetic (PK) parameters were assessed in a sub-group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 2 to 75 years
* Subjects with primary humoral immunodeficiency, namely with a diagnosis of: CVID (Common Variable Immunodeficiency) as defined by PAGID (Pan-American Group for Immunodeficiency) and ESID (European Society for Immunodeficiencies) or XLA (X-linked Agammaglobulinemia)
* Written informed consent

Exclusion Criteria:

* Newly diagnosed PID
* Evidence of an active serious infection at the time of screening (i.e., but not limited to: bacteremia/septicemia, pneumonia, fungal osteomyelitis)
* Malignancies of lymphoid cells such as lymphocytic leukemia, Non-Hodgkin's lymphoma and immunodeficiency with thymoma
* Known hyperprolinemia
* Hypoalbuminemia, protein-losing enteropathies, and any proteinuria
* Allergic reactions to immunoglobulins or other blood products
* Known antibodies to Immunoglobulin A (IgA)
* The subject is receiving steroids (oral and parenteral, daily ≥ 0.15 mg of prednisone equivalent/kg/day) or other systemic immunosuppressants
* Female who is pregnant, breast feeding or planning a pregnancy during the course of the study
* Participation in a study with an investigational product other than (IVIG) within 1 month prior to enrollment
* A positive result at screening on any of the following viral markers: Human Immunodeficiency Virus (HIV), Hepatitis C virus (HCV) and Hepatitis B virus (HBV)
* Aspartate aminotransferase (ASAT) or Alanine aminotransferase (ALAT) concentration > 2.5 times the upper normal limit (UNL)
* Creatinine concentration > 1.5 times the UNL
* Any condition that is likely to interfere with evaluation of the study drug or satisfactory conduct of the trial

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Wasserman, MD, PhD, Principal Investigator — Dallas Allergy Immunology and Medical City Children's Hospital,
Locations (12):
- United States (12):
  - Study Site, Los Angeles, California
  - Study Site, Centennial, Colorado
  - Study Site, North Palm Beach, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Fort Wayne, Indiana
  - Study Site, Indianapolis, Indiana
  - Study Site, Iowa City, Iowa
  - Study Site, St Louis, Missouri
  - Study Site, Newark, New Jersey
  - Study Site, New York, New York
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Dallas, Texas

REFERENCES:
- [Result] Hagan JB, Fasano MB, Spector S, Wasserman RL, Melamed I, Rojavin MA, Zenker O, Orange JS. Efficacy and safety of a new 20% immunoglobulin preparation for subcutaneous administration, IgPro20, in patients with primary immunodeficiency. J Clin Immunol. 2010 Sep;30(5):734-45. doi: 10.1007/s10875-010-9423-4. Epub 2010 May 8. PMID 20454851
- [Result] Wasserman RL, Melamed I, Nelson RP Jr, Knutsen AP, Fasano MB, Stein MR, Rojavin MA, Church JA. Pharmacokinetics of subcutaneous IgPro20 in patients with primary immunodeficiency. Clin Pharmacokinet. 2011 Jun;50(6):405-14. doi: 10.2165/11587030-000000000-00000. PMID 21553933
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20454851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 centers in the United States enrolled subjects for this study.
Groups:
- IgPro20: IgPro20 is a liquid formulation of normal human IgG at a concentration of 20% administered as a SC infusion at weekly intervals.
Period: Wash in/Wash Out Period
Arm/Group | IgPro20
Started | 49
Completed | 38
Not Completed | 11
Not completed — Withdrawal by Subject | 8
Not completed — Adverse Event | 2
Not completed — Disqualifying laboratory results | 1
Period: Efficacy Period
Arm/Group | IgPro20
Started | 38
Completed | 28
Not Completed | 10
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance | 1
Not completed — Termination of study site | 1

BASELINE CHARACTERISTICS:
Arm/Group | IgPro20
Number analyzed (Participants) | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 34.4 (20.09)
Age, Customized [Number; unit: participants]
  2 to < 12 years | 3
  12 to < 16 years | 7
  16 to < 65 years | 33
  ≥ 65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3
  White | 46
Type of Primary Immunodeficiency [Number; unit: participants]
  Common variable immunodeficiency (CVID) | 46 (21.24)
  X-linked agammaglobulinemia (XLA) | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Clinically Documented Serious Bacterial Infections (SBIs) (MITT Population)
Description: The annualized rate was based on the total number of SBIs and the total number of subject study days during the efficacy period for all subjects in the specified analysis population and adjusted to 365 days.
  Potential SBIs included pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess. If an adverse event (AE) was identified as a potential SBI, the AE was adjudicated by a review committee to determine if the event fulfilled the predefined criteria for SBIs.
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: The modified intention-to-treat (MITT) population included all subjects who were treated with IgPro20 during the efficacy period (starting with Week 13) who had the disease under study.
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Efficacy Period Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
Number analyzed (Efficacy Period Subject Study Days) | 12697
SBIs per subject year | 0.00

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) of Total Serum Immunoglobulin G (IgG)
Description: Evaluate non-inferiority of steady-state IgG area under the concentration-time curves standardized to a 7-day period (sAUCs) for subcutaneous immunoglobulin (SCIG) (IgPro20) versus the sAUC under intravenous immunoglobulin (IVIG) (Privigen) treatment. The sAUC under IVIG was taken from the same subjects in a preceding study (either ZLB03_002CR [NCT00168025] or ZLB05_006CR [NCT00322556]).
Time Frame: Measured during a single dosing interval after at least 12 weeks of stable subcutaneous (SC) dosing with IgPro20 treatment
Population: The Per Protocol Pharmacokinetic (PPK) population included all subjects with the disease under study who fulfilled the requirements of the PK substudy, including PK sampling in a preceding study with IVIG (Privigen, CSL Behring), and fulfilling IgPro20 dosing requirements and providing adequate PK blood samples in the current study.
Measure: Mean (Standard Deviation); unit: days*g/L
Groups:
- IgPro20 (PK Substudy): IgPro20 is a liquid formulation of normal human IgG at a concentration of 20% administered as a SC infusion at weekly intervals.
- IVIG (Privigen; Previous Study): Privigen is a liquid formulation of normal human IgG at a concentration of 10% administered as an intravenous infusion every 3 or 4 weeks.
Arm/Group | IgPro20 (PK Substudy) | IVIG (Privigen; Previous Study)
Number analyzed (Participants) | 18 | 18
days*g/L | 105.6 (31.56) | 103.2 (20.00)
Statistical Analysis 1: Comparison: IgPro20 (PK Substudy) vs IVIG (Privigen; Previous Study); Individual sAUC values (standardized to a 7-day period) of the IV and adjusted SC sampling periods in each individual subject were log transformed and a parametric 2-sided 90% confidence interval (CI) for the mean of the individual differences was obtained. Back-transformation of the mean and its CI produced the geometric mean ratio (GMR) and its respective 90% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority of SCIG:IVIG treatment was concluded if the lower GMR confidence limit was 0.8 or more. With 18 evaluable subjects, the power to show this non-inferiority was calculated to be 85% based on the assumptions of an intra-individual variability with a coefficient of variation (CV) = 25% and a GMR equal to or greater than 1; t-test, 2 sided — No P-value is provided as non-inferiority was assessed by the CI of the GMR; Based on log-transformed individual differences; Geometric mean ratio (GMR) = 1.002, 90% CI 2-sided [0.951 to 1.055] — Geometric mean ratio SCIG:IVIG non-inferiority was concluded if the lower GMR confidence limit was 0.8 or more

3. Secondary Outcome: Annualized Rate of Clinically Documented SBIs (ITT Population)
Description: The annualized rate was based on the total number of SBIs and the total number of subject study days during the study for all subjects in the specified analysis population and adjusted to 365 days.
  Potential SBIs included pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess. If an AE was identified as a potential SBI, the AE was adjudicated by a review committee to determine if the event fulfilled the predefined criteria for SBIs.
Time Frame: For the duration of the study, up to 15 months
Population: The Intention To Treat (ITT) population included all subjects who were treated with IgPro20 during any study period.
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 49
Number analyzed (Subject Study Days) | 16234
SBIs per subject year | 0.00

4. Secondary Outcome: Annualized Rate of Clinically Documented SBIs (PPE Population)
Description: The annualized rate was based on the total number of SBIs and the total number of subject study days during the efficacy period for all subjects in the specified analysis population and adjusted to 365 days.
  Potential SBIs included pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess. If an AE was identified as a potential SBI, the AE was adjudicated by a review committee to determine if the event fulfilled the predefined criteria for SBIs.
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: The Per Protocol Efficacy (PPE) population included all subjects who completed the 12-month efficacy period according to the protocol-defined requirements.
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Efficacy Period Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 25
Number analyzed (Efficacy Period Subject Study Days) | 9543
SBIs per subject year | 0.00

5. Secondary Outcome: Annualized Rate of Infection Episodes
Description: The annualized rate was based on the total number of infection episodes occurring during the efficacy period (N = 96) divided by the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: Efficacy period: up to 12 months (week 13 to completion visit)
Population: The MITT population included all subjects who were treated with IgPro20 during the efficacy period (starting with Week 13) who had the disease under study.
Measure: Number (95% Confidence Interval); unit: infection episodes per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
Number analyzed (Subject Study Days) | 12697
infection episodes per subject year | 2.76 [2.235 to 3.370]

6. Secondary Outcome: Number of Infection Episodes (Serious and Non-serious)
Description: Total number of infections for the specified analysis population
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: as for outcome 5
Measure: Number; unit: infections
Arm/Group | IgPro20
Number analyzed (Participants) | 38
infections | 96

7. Secondary Outcome: Annualized Rate of Days Out of Work / School / Kindergarten / Day Care or Unable to Perform Normal Daily Activities Due to Infections
Description: The annualized rate was based on the total number of days out of work / school / kindergarten / day care or inability to perform normal activities due to infection (N = 71), and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: as for outcome 1
Measure: Number; unit: days per subject year
Units Other Than Participants: Exposure Days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
Number analyzed (Exposure Days) | 12605
days per subject year | 2.06

8. Secondary Outcome: Number of Days Out of Work / School / Kindergarten / Day Care or Unable to Perform Normal Daily Activities Due to Infections
Description: Total number of days out of work / school / kindergarten / day care or unable to perform normal daily activities due to infections, for the specified analysis population
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: as for outcome 5
Measure: Number; unit: days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
days | 71

9. Secondary Outcome: Annualized Rate of Hospitalization Due to Infection
Description: The annualized rate was based on the total number of days of hospitalization due to infection (N = 7) and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: as for outcome 5
Measure: Number; unit: days per subject year
Units Other Than Participants: Exposure Days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
Number analyzed (Exposure Days) | 12605
days per subject year | 0.20 [0 to 7]

10. Secondary Outcome: Number of Days of Hospitalization Due to Infections
Description: Total number of days of hospitalization due to infections for the specified analysis population
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: as for outcome 5
Measure: Number; unit: days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
days | 7

11. Secondary Outcome: Use of Antibiotics for Infection Prophylaxis and Treatment
Description: Annualized rate of days with antibiotics for infection prophylaxis and treatment. The annualized rate was based on the total number of days of antibiotic use for infection prophylaxis and treatment in the efficacy period, and the total number of subject study days for all subjects in the specified analysis population, and adjusted to 365 days.
Time Frame: Efficacy period: up to 12 months (week 13 to the completion visit)
Population: as for outcome 5
Measure: Number; unit: days per subject year
Units Other Than Participants: Exposure Days
Arm/Group | IgPro20
Number analyzed (Participants) | 38
Number analyzed (Exposure Days) | 12697
days per subject year | 48.52

12. Secondary Outcome: Total Serum IgG Trough Levels
Description: The IgG trough values per subject were aggregated to a median value, and then median values across subjects were summarized using descriptive statistics.
Time Frame: Every 4 weeks, throughout the 12-month efficacy period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | IgPro20
Number analyzed (Participants) | 38
g/L | 12.53 (3.21)

13. Secondary Outcome: Maximum Concentration (Cmax) of Total Serum IgG at Steady State
Time Frame: Week 28 ± 1 week of the treatment period
Population: The PPK population included all subjects with the disease under study who fulfilled the requirements of the PK substudy, including PK sampling in a preceding study with IVIG (Privigen, CSL Behring), and fulfilling IgPro20 dosing requirements and providing adequate PK blood samples in the current study.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 18
g/L | 16.16 (4.93)

14. Secondary Outcome: Tmax at Steady State
Description: Timepoint of maximum concentration (Cmax)
Time Frame: Week 28 ± 1 week of the treatment period
Population: as for outcome 13
Measure: Median (Full Range); unit: days
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 18
days | 3.118 (1.7729) [0 to 6.97]

15. Other Pre Specified Outcome: Minimum Concentration (Cmin) of Total Serum IgG at Steady State
Time Frame: Week 28 ± 1 week of the treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 18
g/L | 13.70 (4.39)

16. Other Pre Specified Outcome: Rate of All AEs by Relatedness and Seriousness
Description: The rate of AEs was the number of AEs over the number of infusions administered. At least possibly related AEs included possibly related AEs, probably related AEs, and related AEs.
Time Frame: For the duration of the study, up to 15 months
Population: The ITT population included all subjects who were treated with IgPro20 during any study period.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 49
Number analyzed (Infusions) | 2264
AEs per infusion
  All | 0.773
  At least possibly related | 0.634
  Serious | 0.004
  At least possibly related and serious | 0

17. Other Pre Specified Outcome: Rate of Mild, Moderate, or Severe Local Reactions
Description: In addition to the standard MedDRA System Organ Class (SOC) AE assignments, the category of 'local reactions' was defined to provide the possibility for a combined analysis of local reactions and included AEs of injection site reaction, injection site bruising, infusion site scab, injection site cyst, injection site eczema, injection site irritation, injection site nodule, and injection site pain.
  Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
Time Frame: For the duration of the study, up to 15 months
Population: The ITT population included all subjects who were treated with IgPro20 during any study period.
Measure: Number; unit: local reactions per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 49
Number analyzed (Infusions) | 2264
local reactions per infusion
  All | 0.592
  Mild | 0.553
  Moderate | 0.038
  Severe | 0.002

ADVERSE EVENTS:
Time Frame: Approximately 15 months (including the 3 month wash in/wash out period and the 12 month efficacy period).
Description: For the serious AEs (SAEs), treatment-emergent SAEs are provided.
Arm/Group | IgPro20
Serious Adverse Events (participants affected / at risk) | 7/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=49)
Gastroenteritis (Infections and infestations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=49)
Injection site reaction (General disorders) | 49 (1314)
Sinusitis (Infections and infestations) | 14 (20)
Headache (Nervous system disorders) | 13 (40)
Nasopharyngitis (Infections and infestations) | 11 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 7 (8)
Bronchitis (Infections and infestations) | 6 (9)
Fatigue (General disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Acute sinusitis (Infections and infestations) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (11)
Injection site bruising (General disorders) | 5 (19)
Nausea (Gastrointestinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Migraine (Nervous system disorders) | 4 (5)
Pain (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Urinary tract infection (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 4 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Conjunctivitis (Eye disorders) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Influenza (Infections and infestations) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Otitis media (Infections and infestations) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requests that reports based on single-site data not precede the primary publication of the entire clinical trial.